CLINICAL TRIAL: NCT04713462
Title: Real-world Data and Economic Evaluation of Nivolumab in Previously Treated NSCLC Patients in Greece
Brief Title: Real-world Data of Nivolumab in Pre-treated NSCLC
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: HΕ 2B/16
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nivolumab is an approved treatment option for patients with previously treated advanced NSCLC, based on the survival benefit shown versus docetaxel in randomized phase III trials in second line. However, the profile of treatment and even patient outcomes are often different in routine clinical practice than in a clinical trial setting. Furthermore, the financial impact of an approved therapy is often largely unknown. This study will record the efficacy and tolerability of Nivolumab in previously treated patients with NSCLC and describe the treatment patterns and economic impact in real-world settings in Greece.

DETAILED DESCRIPTION:
Patients with advanced NSCLC who had received nivolumab as 2nd line and beyond, between October 2015 and November 2019, in HeCOG clinical centres in Greece, were enrolled. Information regarding detailed patient and treatment characteristics including post-nivolumab therapies, efficacy, and safety data of nivolumab treatment and additionally data on costs and other economic values are collected, analysed and compared with historical data in order to describe the real-world patterns of Nivolumab use in 2nd line NSCLC therapy in Greece.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of advanced Squamous or Non-Squamous NSCLC (histologically or cytologically confirmed), who had relapsed after 1 prior platinum-based systemic treatment and who received treatment with nivolumab
* nivolumab treatment received in participating HeCOG centres between October 2015 and November 2019
* Alive patients must have signed and dated the study approved written informed consent form in accordance with regulatory and institutional guidelines, obtained before any protocol-related procedures that are not part of normal patient care.

Exclusion Criteria:

* Alive patients who do not want to sign and date the study approved written informed consent form
* Patients that participated in any other clinical trial prior or after nivolumab treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced NSCLC who had received nivolumab as 2nd line and beyond, between October 2015 and November 2019, in HeCOG clinical centres in Greece, were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Description of real world clinical use of Nivolumab in pre-treated NSCLC patients | approximately 12 months
  Real-world clinical use
overall survival (OS) | approximately 12 months
  Measured from time of initial treatment with nivolumab until date of death

SECONDARY OUTCOMES:
Objective Response Rate (ORR) as assessed by investigator | approximately 12 months
  the number of participants with best overall response (OR) of confirmed complete response (CR) or partial response (PR) divided by the total number of participants who received treatment
Cost-effectiveness | approximately 12 months
  economic evaluations based on costs of Nivolumab clinical use in Greece

IPD SHARING:
Plan to Share IPD: Undecided